CLINICAL TRIAL: NCT04367090
Title: An Open, Single-arm and Multi-center Pharmacokinetic Study of Pyrotinib and Docetaxel Plus Trastuzumab in Patients With HER2 Positive Recurrent or Metastasis Breast Cancer.
Brief Title: Pharmacokinetic Study of Pyrotinib and Docetaxel in Combination With Trastuzumab in Patients With HER2 Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLTN-Ig
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Trastuzumab; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib and docetaxel plus trastuzumab (Experimental)
  Interventions: Drug: Docetaxel, trastuzumab; Drug: Pyrotinib

INTERVENTIONS:
Drug: Docetaxel, trastuzumab — Docetaxel and trastuzumab once per cycle
Drug: Pyrotinib — Pyrotinib 400/320 mg orally daily

SUMMARY:
The primary objective of the study is to study the pharmacokinetics of pyrotinib and docetaxel plus Trastuzumab in HER2 Positive MBC.

The secondary objective of the study is to evaluate the safety and efficacy (ORR) of pyrotinib and docetaxel plus Trastuzumab in HER2 Positive MBC.

ELIGIBILITY:
Inclusion Criteria:

1. HER2 positive recurrent or metastasis breast cancer.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
3. Adequate organ function.
4. Signed, written inform consent obtained prior to any study procedure.

Exclusion Criteria:

1. Patients received more than 1 line of chemotherapy or immunotherapy in the phase of recurrence / metastasis.
2. History of HER tyrosine kinase inhibitors or monoclonal antibody for breast cancer in any treatment setting，except trastuzumab ,or Pertuzumab used in the neo-adjuvant or adjuvant setting.
3. Assessed by the investigator to be unable receive systemic chemotherapy.
4. History of other malignancy within the last 5 years，except for carcinoma in situ of cervix，basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent.
5. Pregnant or lactating women，or for women of childbearing potential unwilling to use a highly-effective contraception during of the study treatment and for at least 7 months after the last dose of study treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Cmax of pyrotinib and docetaxel | Approximately 2 months
  Peak Plasma Concentration (Cmax) of pyrotinib
Pharmacokinetic parameter: AUC of pyrotinib and docetaxel | Approximately 2 months
  Area under the plasma concentration versus time curve (AUC) of pyrotinib and docetaxel

SECONDARY OUTCOMES:
ORR | Approximately 17 months
  Objective Response Rate
AEs+SAEs | Approximately 17 months
  Adverse Events and Serious Adverse Events
λz | Approximately 6 months
The incidence of≥3 grade diarrhea with different treatment | Approximately 17 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dai L, Gao T, Guo R, Chen Y, Wang J, Zhou S, Tang Y, Chen D, Huang S. Efficacy and safety of pyrotinib-based regimens in HER2 positive metastatic breast cancer: A retrospective real-world data study. Neoplasia. 2024 Oct;56:101029. doi: 10.1016/j.neo.2024.101029. Epub 2024 Jul 17. PMID 39024777